CLINICAL TRIAL: NCT02238002
Title: To Investigate Changes in Anterior Chamber Angle Configuration After Phacoemulsification
Brief Title: Assessment Of Anterior Chamber Configuration Changes After Phacoemulsification
Acronym: AOACCCAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zheng Qian (Other)
Responsible Party: Sponsor-Investigator, Zheng Qian, Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: WZMC2013QQFYJ
Record Dates: First submitted 2014-08-28; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Cataract; Shallow Anterior Chamber; Narrow Angle
Keywords: shallow anterior chamber; narrow angle; SS-OCT
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal angle: normal anterior chamber and open angle eyes underwent cataract surgery
  Interventions: Procedure: cataract surgery
- narrow angle: shallow anterior chamber and narrow angle eyes underwent cataract surgery
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — The patients of both groups underwent cataract surgery

SUMMARY:
To investigate changes in anterior chamber angle configuration after phacoemulsification and intraocular lens (IOL) implantation with Swept-Source Optical Coherence Tomography (SS-OCT).

DETAILED DESCRIPTION:
To investigate changes in anterior chamber angle configuration after phacoemulsification and intraocular lens (IOL) implantation in eyes with a shallow anterior chamber and narrow angle, compared with the eyes with normal anterior chamber and open angle using Swept-Source Optical Coherence Tomography (SS-OCT).

ELIGIBILITY:
Inclusion Criteria:

ACD was less than 2.68mm. the anterior chamber angle width on gonioscopy≤Shaffer 2 .

Exclusion Criteria:

primary or secondary glaucoma, peripheral anterior synechiae, history of ocular surgeries

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who underwent phacoemulsification surgery in Eye Hospital of Wenzhou Medical University
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
anterior chamber angle parameters increased | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yun e Zhao, MD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China